CLINICAL TRIAL: NCT01910961
Title: Impact of Limb Remote Ischemic Preconditioning on Mortality, Hospitalization Costs and Quality of Life During Elective Abdominal Aortic Aneurysm Repair: a Randomized Controlled Trial
Brief Title: Impact of Limb Remote Ischemic Preconditioning on Mortality and Quality of Life During Abdominal Aortic Aneurysm Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cai Li (Other)
Collaborators: Huazhong University of Science and Technology (Other); West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Cai Li, MD, PhD, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LRIP; Liu Kexuan (Other Grant/Funding Number: from National Natural Science Foundation, Beijing, China)
Record Dates: First submitted 2013-06-27; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- limb RIPC (Experimental): limb RIPC protocol was applied after anesthetic induction and before the start of surgery. The limb RIPC was induced by placing a blood pressure cuff on the left upper arm of patient for three inflating-deflating cycles: 5 min inflating to 200 mmHg followed by a 5 min reperfusion with deflating the cuff.
  Interventions: Procedure: limb RIPC
- convention (No Intervention): Adult patients undergoing elective open abdominal aortic aneurysm repair received no treatment after induction of anaesthesia.The control group had an uninflated cuff placed on the left upper arm for 30 min.

INTERVENTIONS:
Procedure: limb RIPC — LRIP consisted of three cycles of left upper limb ischemia induced by inflating a blood pressure cuff on the left upper arm to 200mmHg, with an intervening 5 minutes of reperfusion, during which time the cuff was deflated
  Other Names: limb remote ischemic preconditioning
  Arms: limb RIPC

SUMMARY:
To investigate the influence of limb remote ischemic preconditioning (LRIP) on mortality, hospitalization costs and quality of life in patients undergoing open infrarenal abdominal aortic aneurysm (AAA) repair.

DETAILED DESCRIPTION:
Remote ischaemic preconditioning may confer the cytoprotection in critical organs. The investigators have revealed that limb remote ischemic preconditioning (RIPC) would reduce intestinal and pulmonary injury in patients undergoing open infrarenal abdominal aortic aneurysm (AAA) repair.Few groups have investigated the long term influence of limb remote ischemic preconditioning.Therefore, the investigators evaluated the impact of limb remote ischemic preconditioning on mortality, hospitalization costs and quality of life during elective abdominal aortic aneurysm repair in a prospective, randomized, controlled, single blind setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of abdominal aortic aneurysm
* Must be received open abdominal aortic aneurysm repair

Exclusion Criteria:

* age >80 years old
* Acute coronary syndrome or myocardial infraction within 3 months
* Chronic obstructive pulmonary emphysema
* angina pain within 48 hours of repair procedure
* ejection fraction less than 40%
* poor pulmonary function (PaO2 <60mmHg)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

SECONDARY OUTCOMES:
hospitalization costs | 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Kexuan Liu, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250